CLINICAL TRIAL: NCT00739453
Title: A Phase I Dose-escalation Study of OSI-906 and Erlotinib (Tarceva®) in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Dose-escalation Study of OSI-906 and Erlotinib (Tarceva®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-906-103; 2008-001743-20 (EudraCT Number)
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Pancreatic cancer; Advanced cancer; Prostate cancer; Non-small cell lung cancer; Colorectal cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Schedule 1 (Experimental): OSI-906 is administered on Days 1-3 every 7 days. Erlotinib will be administered daily starting on Day 2 of the initial treatment period and on Day 1-21 for all remaining treatment periods.
  Interventions: Drug: OSI-906; Drug: erlotinib
- Schedule 2 (Experimental): OSI-906 is administered daily starting on Day 1 and erlotinib is administered daily starting on Day 2 of the initial treatment period and on Day 1-21 for all remaining treatment periods.
  Interventions: Drug: OSI-906; Drug: erlotinib
- Schedule 3 (Experimental): OSI-906 is administered continuously twice daily starting on Day 1 and erlotinib is administered daily starting on Day 2. The NSCLC expansion cohort will follow Schedule 3 with the exception that erlotinib is administered daily starting on Day 8.
  Interventions: Drug: OSI-906; Drug: erlotinib

INTERVENTIONS:
Drug: OSI-906 — administered orally
Drug: erlotinib — administered orally
  Other Names: Tarceva; OSI-774

SUMMARY:
Multicenter, open-label, phase 1, cohort dose escalation study to determine the Maximum Tolerated Dose (MTD) of OSI-906 in combination with erlotinib

DETAILED DESCRIPTION:
The study will open with Schedule 1 (S1), in which OSI-906 is administered on Days 1-3 every 7 days. Erlotinib will be administered daily starting on Day 2. A treatment period is defined as 21 days.

Initiation of Schedule 2 (S2), in which OSI-906 is administered daily starting on Day 1 and erlotinib is administered daily starting on Day 2, will occur after observation of clinically significant related toxicity >/= grade 2 in any patient on S1 or after > 2 dose levels in S1 have been examined without evidence of Dose Limiting Toxicities (DLT).

Initiation of Schedule 3 (S3), in which OSI-906 is administered twice daily starting on Day 1 and erlotinib is administered daily starting on Day 2, will occur after observation of clinically significant related toxicity >/= grade 2 in any patient on S2 or after > 2 dose levels in S2 have been examined without evidence of DLT.

Once the phase 2 dose has been established for S3, 1 expansion cohort will be opened.

The Expansion Cohort will enroll approximately 30 evaluable patients with stage IIIB/IV Non-small Cell Lung Carcinoma (NSCLC). Patients in the NSCLC Expansion Cohort will be required to have either archival tissue or fresh tumor tissue available at the start of study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumor
* For the NSCLC Expansion Cohort, a confirmed diagnosis of stage IIIB/IV NSCLC after failure of at least 1 prior chemotherapy regimen is required
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status </= 2
* Predicted life expectancy >/= 12 weeks
* Patients may have had prior therapy, providing certain conditions are met:

  1. Chemotherapy: A minimum of 3 weeks (4 weeks for carboplatin or investigational anticancer agents and 6 weeks for nitrosoureas and mitomycin C) must have elapsed between the end of treatment and registration into this study. Patients must have recovered from any treatment-related toxicities (except for alopecia, fatigue, and grade 1 neurotoxicity) prior to registration.
  2. Hormonal therapy: Patients may have had prior anticancer hormonal therapy provided it is discontinued prior to registration into the study. However, patients with prostate cancer with evidence of progressive disease may continue on therapy that produces medical castration (eg, goserelin or leuprorelin), provided this therapy was commenced at least 3 months earlier.
  3. Radiation: Patients may have had prior radiation therapy provided they have recovered from the acute, toxic effects of radiotherapy prior to registration. A minimum of 21 days must have elapsed between the end of radiotherapy and registration into the study unless the radiation affected less than 25% of bone marrow.
  4. Surgery: Previous surgery is permitted provided that wound healing has occurred prior to registration.
* Fasting glucose </= 125 mg/dL (7 mmol/L) at baseline and on Day 1 prior to dosing
* Blood ketones </= Upper Limit of Normal (ULN)
* Neutrophil count >/= 1.5 x 10^9/L
* Platelets >/= 100 x 10^9/L
* Bilirubin </= 1.5 x ULN
* AST and/or ALT </= 2.5 x ULN or </= 5 x ULN if patient has documented liver metastases
* Serum creatinine </= 1.5 x ULN
* Patients must be nonsmokers (or former smokers who stopped smoking > 3 months previously) and have a negative cotinine test at baseline and on Day 1
* Patients in the NSCLC Expansion Cohort must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients in the NSCLC Expansion Cohort will be required to have either an archival or fresh tumor tissue (whole or partial block) available at the start of study
* Patients must be accessible for repeat dosing and follow-up, including pharmacokinetic sampling
* Patients - both males and females - with reproductive potential must agree to practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test at baseline and on Day 1
* Patients must provide verbal and written informed consent to participate in the study

Exclusion Criteria:

* Documented history of diabetes mellitus
* History of significant cardiac disease unless the disease is well-controlled. Significant cardiac diseases includes second/third degree heart block; significant ischemic heart disease; QTc interval > 450 msec at baseline; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea)
* History of cerebrovascular accident (CVA) within 12 months prior to registration or that is not stable
* Prior epidermal growth factor receptor (EGFR) or insulin like growth factor receptor (IGFR) inhibitor therapy, except for prior erlotinib therapy in the NSCLC Expansion Cohort, prior erlotinib therapy will not be exclusionary
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnant or breast-feeding females
* Gastrointestinal (GI) abnormalities including inability to take oral medication, requirement for intravenous (IV) alimentation, active peptic ulcer, or prior surgical procedures affecting absorption
* Ocular inflammatory or infectious condition that is not completely resolved prior to registration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug
* Any type of active seizure disorder
* Use of drugs that have a risk of causing QT interval prolongation within 14 days prior to Day 1 dosing
* Use of strong or moderate CYP3A4 or CYP1A2 inhibitors/inducers, with the exception of low-dose steroids, within 14 days prior to Day 1 dosing
* Use of proton pump inhibitors within 14 days prior to day 1 dosing
* Symptomatic brain metastases that are not stable, require steroids, or that have required radiation within the last 28 days
* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's ongoing participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-10-23 (Actual); Primary Completion 2012-03-03 (Actual); Study Completion 2012-03-03 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and recommended phase 2 dose of OSI-906 and erlotinib | 21 days

SECONDARY OUTCOMES:
Safety profile, Pharmacokinetic profile, pharmacodynamic activity, Preliminary antitumor activity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director, Study Director — Astellas Pharma Global Development
Locations (4):
- United States (3):
  - University of Colorado Health Science Center, Aurora, Colorado
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Hudson-Webber Cancer Research Center, Karmanos Cancer Institute, Detroit, Michigan
- University of Oxford Department of Medical Oncology, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=271